CLINICAL TRIAL: NCT01704846
Title: Assessment of Bioequivalence Between Two Different Formulations of BI 201335 NA Soft Gelatine Capsules in Healthy Male Volunteers. (an Open-label, Randomised, Single-dose, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence Trial of 2 Dose Strengths of BI 201335 NA Soft Gelatine Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1220.53
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

ARMS (2):
- Treatment sequence 1 (Experimental): Test - Reference - Reference - Test
  Interventions: Drug: BI 201335 NA 120 mg capsule; Drug: BI 201335 NA 40 mg capsule
- Treatment sequence 2 (Experimental): Reference - Test - Test - Reference
  Interventions: Drug: BI 201335 NA 120 mg capsule; Drug: BI 201335 NA 40 mg capsule

INTERVENTIONS:
Drug: BI 201335 NA 120 mg capsule — 1capsule of BI 201335 NA 120 mg capsule
  Arms: Treatment sequence 2
Drug: BI 201335 NA 120 mg capsule — 1 capsule of BI 201335 NA 120 mg capsule
  Arms: Treatment sequence 1
Drug: BI 201335 NA 40 mg capsule — 3 capsules of BI 201335 NA 40 mg capsule
  Arms: Treatment sequence 1
Drug: BI 201335 NA 40 mg capsule — 3 capsules of BI 201335 NA 40 mg capsule
  Arms: Treatment sequence 2

SUMMARY:
The objective is to investigate the bioequivalence of 2 dose strengths of 40 mg and 120 mg BI 201335 NA soft gelatine capsules.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male volunteers without any clinical significant findings and complications
2. Age: 20 - 45 years
3. BMI: 18.5 - 25.0 kg/m2
4. Signed informed consent

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance.
2. Any evidence of a clinically relevant concomitant disease according to investigator's clinical judgement.
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
4. History of jaundice
5. Surgery of the gastrointestinal tract (except appendectomy).
6. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
7. History of relevant orthostatic hypotension, fainting spells or blackouts.
8. Chronic or relevant acute infections.
9. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients) according to investigator's clinical judgement.
10. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
11. Use of drugs which might reasonably influence the results (pharmacokinetic) of the trial within at least 10 days prior to administration or during the trial.
12. Participation in another trial with an investigational drug within two months prior to administration or during the trial.
13. Smoking (>10 cigarettes or >3 cigars or >3 pipes/day).
14. Inability to refrain from smoking during the trial.
15. Alcohol abuse (more than 60 g/day: e.g., 3 middle-sized bottles of beer, 3 gous [equivalent to 540 mL] of sake).
16. Drug abuse.
17. Blood donation (more than 100 mL within four weeks prior to administration).
18. Excessive physical activities (within one week prior to administration).
19. Any laboratory value outside the reference range that is of clinical relevance according to investigator's clinical judgement.
20. Any history of relevant liver diseases (for instance, disturbances of liver function, Dubin-Johnson syndrome, Rotor syndrome, or previous liver tumours).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.53.08101 Boehringer Ingelheim Investigational Site, Sumida-ku,Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1: Treatment sequence: Test - Reference - Reference - Test
  Test product: Oral administration of faldaprevir 120 mg (40 mg x 3 soft gelatine capsules) with 150 mL water after an overnight fast.
  Reference Product: Oral administration of faldaprevir 120 mg (120 mg x 1 soft gelatine capsule) with 150 mL water after an overnight fast.
  Treatments were separated by a washout period of at least 14 days.
- Treatment Sequence 2: Treatment sequence: Reference - Test - Test - Reference
  Test product: Oral administration of faldaprevir 120 mg (40 mg x 3 soft gelatine capsules) with 150 mL water after an overnight fast.
  Reference Product: Oral administration of faldaprevir 120 mg (120 mg x 1 soft gelatine capsule) with 150 mL water after an overnight fast.
  Treatments were separated by a washout period of at least 14 days.
Period: Treatment Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 3
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.7) | 30.1 (5.8) | 29.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of the Analyte From Time 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the faldaprevir in plasma over the time interval from 0 to the time of the last quantifiable data point.
  Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: 3 hours (h) before drug administration and 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h and 96h after drug administration
Population: Pharmacokinetic (PK) set included all healthy subjects in the treated set who have evaluable pharmacokinetic variable in the treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Units Other Than Participants: Observations
Groups:
- Test Product: Faldaprevir 40 mg x 3 Capsules: Faldaprevir 120 mg (40 mg x 3 capsules) - soft gelatine capsule- Oral administration with 150 mL water after an overnight fast
- Reference Product: Faldaprevir 120 mg x 1 Capsule: Faldaprevir 120 mg (120 mg x 1 capsules) - soft gelatine capsule- Oral administration with 150 mL water after an overnight fast
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
ng·h/mL | 17297.157 (19.71) | 17216.514 (23.89)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — Assessment of bioequivalence between two different formulations of faldaprevir soft gelatine capsules in healthy male volunteers. The acceptance range for the geometric mean ratio was 80 to 125%; Adjusted Geometric Mean Ratio (%) = 100.47, 90% CI 2-sided [95.90 to 105.25] — Ratio calculated as Test product divided by reference product

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of faldaprevir in plasma. Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
ng/mL | 943.868 (32.16) | 916.480 (39.22)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 102.99, 90% CI 2-sided [95.57 to 110.98] — Ratio calculated as Test product divided by reference product

3. Secondary Outcome: Area Under the Curve Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of faldaprevir in plasma over the time interval from 0 extrapolated to infinity.
  Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
ng*h/mL | 18422.006 (19.07) | 18323.189 (23.18)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 100.54, 90% CI 2-sided [96.10 to 105.18] — Ratio calculated as Test product divided by reference product

4. Secondary Outcome: Time From Dosing to the Maximum Measured Concentration (Tmax)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma.
  Means presented are adjusted means and the standard deviation is actually the intra-individual coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
hours | 4.478 (25.60) [2 to 8] | 4.585 (31.48) [2 to 10]
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — Assessment of bioequivalence between two different formulations of faldaprevir soft gelatine capsules in healthy male volunteers. The acceptance range for the adjusted mean ratio was 80 to 125%; Adjusted Mean Ratio (%) = 97.66, 90% CI 2-sided [91.54 to 103.78] — Ratio calculated as Test product divided by reference product

5. Secondary Outcome: Terminal Rate Constant (λz)
Description: Terminal rate constant of the analyte in plasma. Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
1/h | 0.0265 (9.91) | 0.0264 (6.91)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 100.34, 90% CI 2-sided [98.51 to 102.20] — Ratio calculated as Test product divided by reference product

6. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal half-life of faldaprevir in plasma. Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
hours | 26.204 (9.91) | 26.293 (6.91)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 99.66, 90% CI 2-sided [97.85 to 101.51] — Ratio calculated as Test product divided by reference product

7. Secondary Outcome: Mean Residence Time (MRTpo)
Description: Mean residence time of the analyte in the body after oral administration. Geometric means presented are adjusted means and the coefficient of variation is the intra-individual geometric coefficient of variation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Units Other Than Participants: Observations
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Number analyzed (Participants) | 59 | 60
Number analyzed (Observations) | 118 | 119
hour | 29.948 (9.93) | 29.888 (9.79)
Statistical Analysis 1: Comparison: Test Product: Faldaprevir 40 mg x 3 Capsules vs Reference Product: Faldaprevir 120 mg x 1 Capsule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted Geometric Mean Ratio (%) = 100.20, 90% CI 2-sided [98.10 to 102.34] — Ratio calculated as Test product divided by reference product

ADVERSE EVENTS:
Time Frame: Four treatment periods (Period 1 to 4) of 6 days for each (Days -1 to 5) + Washout period of at least 14 days between treatments
Arm/Group | Test Product: Faldaprevir 40 mg x 3 Capsules | Reference Product: Faldaprevir 120 mg x 1 Capsule
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 7/59 | 8/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product: Faldaprevir 40 mg x 3 Capsules (N=59) | Reference Product: Faldaprevir 120 mg x 1 Capsule (N=60)
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastroenteritis (Gastrointestinal disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.